CLINICAL TRIAL: NCT07390149
Title: The 30-15 Intermittent Fitness Test Provides Superior Sport-Specific Sensitivity to Treadmill Testing in Elite Female Footballers
Brief Title: Fitness Tests Conducted at Intervals of 30-15 Minutes Provide Superior Sport-specific Accuracy Compared to Treadmill Tests in Elite Female Soccer Players.
Acronym: 30-15IFT vs TR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gümüşhane Universıty (Other)
Collaborators: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Coşkun YILMAZ, ASSOC. PROF., Gümüşhane Universıty
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2023/09
Record Dates: First submitted 2026-01-18; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Exercise Physiology; Sports Performance
Keywords: women's football; aerobic capacity; lactate threshold; metabolic response; running performance; intermittent fitness assessment

STUDY DESIGN:
Intervention Model Description: This study used a randomized crossover design in which all participants completed both the 30-15 Intermittent Fitness Test and a treadmill-based incremental running test. The order of the test protocols was randomized, and a 48-hour recovery period was implemented between sessions to minimize carryover effects. Physiological responses were compared within participants across the two testing conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30-15 Intermittent Fitness Test (30-15IFT) (Other): Participants performed the 30-15 Intermittent Fitness Test consisting of 30-second running bouts interspersed with 15-second passive recovery periods, with progressive increases in running speed until volitional exhaustion.
  Interventions: Other: 30-15 Intermittent Fitness Test; Other: Treadmill Incremental Test
- Treadmill Incremental Running Test (TR) (Other): Participants performed a laboratory-based incremental treadmill running test with speed increases every 4 minutes until volitional exhaustion.
  Interventions: Other: 30-15 Intermittent Fitness Test; Other: Treadmill Incremental Test

INTERVENTIONS:
Other: 30-15 Intermittent Fitness Test — Participants performed the 30-15 Intermittent Fitness Test consisting of 30-second running bouts interspersed with 15-second passive recovery periods, with progressive increases in running speed until volitional exhaustion.
Other: Treadmill Incremental Test — Participants performed a laboratory-based incremental treadmill running test with speed increases every 4 minutes until volitional exhaustion.

SUMMARY:
This study compares the acute aerobic, metabolic, and threshold-related physiological responses elicited by the 30-15 Intermittent Fitness Test (30-15IFT) and a treadmill-based incremental running test in elite female football players. Using a randomized crossover design, all participants completed both testing protocols with a 48-hour recovery period. Outcomes included maximal oxygen uptake, maximal running speed, heart rate responses, lactate-derived thresholds, metabolic tolerance indices, and recovery markers.

DETAILED DESCRIPTION:
Laboratory-based treadmill tests are commonly used to assess aerobic capacity in football players; however, they lack sport-specific characteristics such as intermittent running, accelerations, and changes of direction. The 30-15 Intermittent Fitness Test (30-15IFT) has been proposed as a more ecologically valid field-based alternative.

Twenty-seven elite female football players competing in the Turkish Women's Super League completed both the 30-15IFT and a standardized treadmill incremental protocol in a randomized crossover design. Tests were separated by 48 hours and performed under controlled environmental conditions. Physiological variables including VO₂max, maximal running speed, maximal heart rate, respiratory exchange ratio, lactate-derived thresholds (OBLA), metabolic load-dependent tolerance, and post-exercise recovery markers were assessed using breath-by-breath gas analysis, heart rate monitoring, and capillary blood lactate sampling.

The study aims to determine whether the 30-15IFT elicits more sensitive and sport-specific physiological responses compared with treadmill testing, thereby supporting its use in performance monitoring and individualized training prescription in elite women's football.

ELIGIBILITY:
Inclusion Criteria:

* Female football players aged 18-35 years
* Competing in the Turkish Women's Super League
* Minimum of 3 years of professional football experience,
* Full participation in training and matches during the previous 6 months,
* Ability to perform maximal exercise testing

Exclusion Criteria:

* Musculoskeletal injury affecting performance within the last 3 months,
* Diagnosed cardiovascular, metabolic, or respiratory disease,
* Any condition limiting maximal physical effort

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 27 (Actual)
Dates: Start 2025-01-05 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Maximal Oxygen Uptake (VO₂max) | Day 1
  Maximal oxygen uptake measured via breath-by-breath gas analysis.
Maximal Running Speed (MRS) | Day 1
  Highest running speed achieved during each protocol.

SECONDARY OUTCOMES:
Maximal Heart Rate (HRmax) | During exercise
  Peak heart rate achieved during each test.
Respiratory Exchange Ratio (RER) | End of exercise
  Ratio of carbon dioxide production to oxygen uptake.
Onset of Blood Lactate Accumulation (OBLA) | Post-exercise (3 min)
  Running speed, VO₂, and heart rate corresponding to 4 mmol·L-¹ blood lactate.
Maximum Lactate Delayed Time (MLDT) | Post-exercise
  Time from exercise cessation to peak blood lactate concentration.
Blood Lactate Concentration (L3MAT) | post-exercise
  Capillary blood lactate concentration during recovery.
Heart Rate Recovery (HR3AT) | Post-exercise
  Heart rate values during recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Coşkun YILMAZ, associate professor, Study Chair — Gümüşhane Üniversity
Locations (1):
- Gumushane Univetsity, Gümüşhane, Gümüşhane Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset consists of a small sample of elite athletes, and sharing de-identified data could still pose a risk of participant re-identification. In addition, no data-sharing agreement or participant consent for IPD sharing was established at the time of study design. Aggregate data supporting the findings are reported within the published article.